CLINICAL TRIAL: NCT04515758
Title: Combined Cognitive and Exercise Training for Older Adults: Feasibility & Effectiveness
Brief Title: Determining the Feasibility of Implementing a Combined Cognitive and Exercise Training Program for Older Adults in a Community Setting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Royal Bank of Canada (Unknown); YMCA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 40928
Record Dates: First submitted 2020-04-16; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Osteo Arthritis; Osteoporosis; Joint Replacement; Fibromyalgia; High Blood Pressure; Stable Heart Conditions; Chronic Obstructive Pulmonary Disease; Diabetes; Obesity
Keywords: Feasibility; Exercise training; Cognitive Training; Chronic conditions; Older adults; Community setting
MeSH Terms: conditions — Osteoporosis; Fibromyalgia; Hypertension; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Obesity; Chronic Disease | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the exercise only group or the cognitive training and exercise group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are told that there are two intervention groups ("regular exercise group" and an "augmented exercise group"). They are not told how the two group interventions differ (i.e. they are unaware of which group they were assigned to, as they do not know what intervention is being delivered to the other group). Assessors of the outcomes are not aware of which group the participant's have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Cognitive Training (Experimental): Each participant (in a group setting) completes 30 minutes of cognitive training and 1 hour of exercise two days/week.
  Interventions: Other: Exercise and Cognitive Training
- Exercise Training Only (Active Comparator): Each participant (in a group setting) completes 1 hour of exercise two days/week (separate days than the experimental group).
  Interventions: Other: Exercise Training Only

INTERVENTIONS:
Other: Exercise and Cognitive Training — Exercise: 12-week, twice-weekly 60-minute program. Each session includes a brief 5 minute educational lesson on a health-related topic (i.e. healthy eating, good posture, etc.). Each participant receives individualized and progressive exercise program from qualified exercise providers (YMCA instructors). The programs include whole body exercises including squats, rows, chest press, bicep/tricep exercises, shoulder exercises, and core exercises. A 5 warm-up is done (individually or in a group) and a 5 minute group cool-down (stretching) is done each class. Cognitive training: focuses on dual-task training (provided by an Android tablet). Each cognitive task requires the participant to choose and execute the response appropriate for the stimuli presented. Participants must prioritize their response and perform tasks as fast as possible while maintaining accuracy. The difficulty of the training is individualized and progressive based on their ongoing performance.
  Arms: Exercise and Cognitive Training
Other: Exercise Training Only — Exercise: 12-week, twice-weekly 60-minute program. Each session includes a brief 5 minute educational lesson on a health-related topic (i.e. healthy eating, good posture, etc.). Each participant receives individualized and progressive exercise program from qualified exercise providers (YMCA instructors). The programs include whole body exercises including squats, rows, chest press, bicep/tricep exercises, shoulder exercises, and core exercises. A 5 warm-up is done (individually or in a group) and a 5 minute group cool-down (stretching) is done each class.
  Arms: Exercise Training Only

SUMMARY:
The overarching aim of this project is to implement and evaluate a proven cognitive training regimen in combination with a community exercise program among older adults who attend wellness exercise programs at the YMCA. To support this aim, the investigators have developed a collaboration with the YMCA of Kitchener-Waterloo, which offer exercise programs targeted to older adults. The specific objectives are: (1) to evaluate the feasibility of a combined exercise and cognitive training in a community-setting among older adults; and (2) to conduct a preliminary evaluation and comparison of changes in cognitive function, physical function, well-being and self-efficacy with 12-weeks of combined exercise and cognitive training versus exercise alone. The hypothesis for each objective are as follows: (1) It is anticipated that this program will be feasible to implement and will be well accepted by the participants and exercise providers. (2) The investigators may not have the power to find statistically significant differences between the control and experimental groups for physical and cognitive function. However, the investigators expect to observe positive changes between the pre- and post-assessments, suggesting improved cognitive function and mobility as a result of the 12-week program.

DETAILED DESCRIPTION:
The study will be conducted at the A. R. Kaufman YMCA fitness center where 32 registrants of the "Move for Health Program" (formally known as the Live Smart program) will be asked to participate. The "Move for Health" program is a 12-week, twice-weekly 60 minute program that includes both aerobic and strength training. The cognitive training (delivered by an Android Tablet) focuses on dual-task training and requires participants to employ higher-order cognitive abilities such as attention and executive function. 16 Participants in one group will complete cognitive training integrated into the Move for Health exercise program, whereas 16 participants in the other group (completing program on separate days) will complete the exercise program only. All participants will complete assessments of cognitive function, physical function, well-being, and self-efficacy before and after the programs. This study will be the first to examine the feasibility, acceptability, and effectiveness of a combined cognitive and exercise training program for older adults in a community-setting. If shown to be feasible, it has the potential for broader investigation and, eventually, wide-scale implementation to benefits the health of older Canadians.

Note: Due to low recruitment rates, 11 participants were recruited in the Fall of 2019 and all completed the experimental intervention. 32 participants were recruited and randomized for the Winter of 2020. In response to COVID-19, the YMCA shut down and thus the intervention has halted prematurely after 6 weeks of program. Post-program updated demographic information, activity questionnaires (physical, cognitive, and social), and assessments for overall well-being and self-efficacy will be conducted over phone or video call.

ELIGIBILITY:
Inclusion Criteria:

* Must be available and willing to participate during the schedule program days and times (which were determined based on the scheduling of other regular YMCA programs)
* Communicate proficiently in English (i.e. would be able to understand and respond to instructions and questions that provided both verbally and in written form in English)
* Must have one or more of the following chronic conditions: including osteoarthritis, osteoporosis, pre/post-joint replacement, fibromyalgia, high blood pressure, stable heart conditions, Chronic Obstructive Pulmonary Disease, diabetes, and/or obesity.
* When wearing their usual corrective lenses, they are able to read standard newsprint
* While wearing their normal hearing aid (if required), they are able to converse with another person in a public area or somewhat crowded room

Exclusion Criteria:

* Currently undergoing treatment for cancer (not included in this specific YMCA program's target participants)
* Has completed this specific YMCA exercise program within the last year
* Has been diagnosed with a concussion and/or has been experiencing concussion-related symptoms in the last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Pre-program (baseline)
  Total number of people enrolled divided by the total number of people invited to participate (multiplied by 100 to calculate a percentage)
Completion Rate | Through study completion, 12 weeks
  Percentage of people who completed the full program and all assessments
Attendance | Throughout entire intervention (12 weeks, 2 sessions/week per group)
  Percentage of people who attended program sessions (exercise and cognitive training components)
Change in Participant and Instructor Rating of experience, satisfaction, and feasibility of program | Mid-point (6 weeks) and post-program (12 weeks)
  Participant and instructors rating of program components and overall program (via hand-written questionnaire). Participants and instructors must rate their level of agreement (1 = strongly disagree, 2 = disagree, 3 = no opinion, 4 = agree, 5 = strongly agree) with various statements. The higher the rating, the greater the satisfaction. They also must rate if the difficulty of the program was optimal, somewhat easy or hard, or too easy or hard. They must also specify how much money they would be willing to spend on the program. They are also given an opportunity to record optional additional comments/recommendation.
Cost of program | Post-program (12 weeks)
  Financial cost of running program (equipment purchased for study - cognitive training tablet and stands - and YMCA staff pay) as reported by researcher and YMCA staff
Sex | Pre-program (baseline)
  Self-reported biological sex (at birth) using basic demographics questionnaire
Participant and Instructor perceived program experience and satisfaction | Post-program (at 12 weeks)
  One-on-one interview with researcher, answering broad questions about their experience in the program and study
Participant and Instructor observer-perceived program experience and satisfaction | Throughout entire intervention (12 weeks, 2 sessions/week per group)
  Experience of participants and instructors will also be observed by the researcher (observational notes will be taken by the researcher during each class). No names of participants and instructors will be recorded.
Education | Pre-program (baseline)
  Self-reported years of formal education and training (training years for instructors only) using basic demographics questionnaire
Occupation | Pre-program (baseline)
  Self-reported previous and current occupations using basic demographics questionnaire
Medical Condition | Pre-program (baseline)
  Self-reported previous and current medical conditions using basic demographics questionnaire
Medications | Pre-program (baseline)
  Self-reported previous and current medications using basic demographics questionnaire
Montreal Cognitive Assessment (global cognitive function) | Pre-program (baseline)
  Using the Montreal Cognitive Assessments (brief clinical tool) to assess visual/spatial abilities, working memory, executive functioning, language, abstraction, and orientation). Will be used to describe participants' baseline cognitive status (a score out of 30 is measured).
Physical Activity Level | Pre-program (baseline)
  Using the International Physical Activities Questionnaire (IPAQ) to assess physical activity level based on self-reported frequency and duration of job-related, house work-related, transportation-related, and leisure-related physical activities done in the past week. METS-minutes/week will be calculated and reported (i.e. take the number of minutes doing an activity in the past week and multiply by the appropriate metabolic equivalent, which will vary based on the intensity of the physical activity).
Participant cognitive activity | Pre-program (baseline)
  Using a cognitive activity scale (score of 0-4 per activity) that requires participants to self-report how often they typically engage in a variety of mentally stimulating activities (i.e. playing card games, reading, cooking, etc.) The more frequently they engage in the activity, the higher the score.
Participant social activity | Pre-program (baseline)
  Using a scale (score of 0-3 per group) that requires participants to self-report how often they typically interact (face-to-face or virtually) with different groups of people (i.e. their spouse, family, friends, co-workers, etc.). The more frequently they interact with the group, the higher the score.
Participant and Instructor Age | Pre-program (baseline)
  Self-reported years of age using basic demographics questionnaire

SECONDARY OUTCOMES:
Change in Stroop Task Performance | Pre-program (baseline) and post-program (12 weeks)
  STROOP task which assesses the length of time (seconds) it takes for a participant to correctly name a coloured square (test 1), read the name of a colour (test 2), and say the name of the colour that a word is printed in (test 3). Number of corrected and uncorrected errors are also recorded.
Change in Trail Making Task Performance | Pre-program (baseline) and post-program (12 weeks)
  Trails Making Test Part A and B. Part A assesses visual search (participants must connect numbered circles in ascending numerical order (1-2-3-etc). Part B assesses working memory and task-switching (participants must connect circles in ascending numerical and alphabetical order (1-A-2-B- etc.). Time to complete the tests (second) and errors (number) made during the tests are recorded.
Change in Resting Heart Rate | Pre-program (baseline) and post-program (12 weeks)
  Resting (seated) heart rate (beats per minute) using an automatic blood pressure cuff
Change in Resting Systolic and Diastolic Blood Pressure | Pre-program (baseline) and post-program (12 weeks)
  Resting (seated) blood pressure (millimeters of mercury) using an automatic blood pressure cuff
Change in Grip Strength | Pre-program (baseline) and post-program (12 weeks)
  Using hand dynamometer (assessing grip strength in lbs) for right and left hand (two trials per hand)
Change in Body Mass Index (BMI) | Pre-program (baseline) and post-program (12 weeks)
  Weight (using automatic scale to measure in lbs, converted to kg) and height (measured in feet and inches, converted to meters) measured and combined to provide BMI (kg/m^2)
Change in Hip-to-Waist Circumference Ratio | Pre-program (baseline) and post-program (12 weeks)
  Divide waist circumference (cm) by hip circumference (cm) to get ratio calculation
Change in Timed Up-and-Go Performance | Pre-program (baseline) and post-program (12 weeks)
  Agility and functional balance will be assessed using the Timed Up-and-Go (participants stand up from a chair, walk 6 meters, turn around an object, walk back to chair, and sit down). Time to complete test is measured (seconds) and assessor's observational notes of performance are taken.
Change in Four Square Step Test Performance | Pre-program (baseline) and post-program (12 weeks)
  Agility and functional balance will be assessed using the Four Square Step Test (participants must step over lines that are set up in a cross formation, creating 4 quadrants. They must step forward, backward, and side to side in a specific pattern (i.e. from quadrant 1 to quadrant 2, to quadrant 3, to quadrant 4). Time to complete test is recorded in seconds.
Change in Sit-to-Stand Performance | Pre-program (baseline) and post-program (12 weeks)
  Lower body strength will be assessed using the 5 Time Sit-to-Stand (participants must complete 5 sit-to-stands from a chair as fast as they can). Time to complete all 5 is recorded in seconds.
Change in 6-minute walk test Performance | Pre-program (baseline) and post-program (12 weeks)
  Functional fitness will be assessed using the 6 minute walk (participants walk along indoor track for 6 minutes). The number of laps achieved in 6 minutes is recorded. Assessor's observational notes of walking performance is also recorded.
Change in Overall Well-being | Pre-program (baseline) and post-program (12 weeks)
  Well-being will be self-reported using the "Vitality-Plus Scale" (self-reported general health questionnaire - rating of sleep quality, appetite, general energy level, etc.). Participants rate their degree of health on a scale from 1 - 5 (the higher the rating, the better their perceived overall well-being).
Change in Exercise-related Self-Efficacy | Pre-program (baseline) and post-program (12 weeks)
  Bandura Scale (named after the researcher who developed it) - self-reported rating of confidence (0 - 100%) to continue exercising routinely in various hypothetical situations (i.e. if one is sick, if the weather is poor, etc). The greater the confidence, the higher the score

CONTACTS AND LOCATIONS:
Locations (1):
- A. R. Kaufman YMCA, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No